CLINICAL TRIAL: NCT02518022
Title: A Monocentric, Controlled, Randomized, Open-label Cross-over Study to Explore the Possible Insulin Treatment of Beverages Containing Alcohol and Carbohydrates in Adolescents and Young Adults With Type 1 Diabetes
Brief Title: How to be Safe With Alcoholic Drinks in Diabetes
Acronym: BEER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unexpected low willingness of patient to participate on the study
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BEER2015
Record Dates: First submitted 2015-05-22; First posted 2015-08-07 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
Keywords: Type 1 Diabetes mellitus; Hypoglycemia; continuous subcutaneous insulin infusion; Alcohol; continuous glucose monitoring system; Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Insulin; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): For carbohydrates in beer, subjects will get covering by Insulin (1/2 of calculated amount). As well Insulin basal rate will set to half for 12 hours
  Interventions: Drug: Insulin
- Standard (No Intervention): No Insulin Treatment of carbohydrates in beer.

INTERVENTIONS:
Drug: Insulin — Insulin for beer
  Other Names: Novorapid or Humalog
  Arms: Intervention

SUMMARY:
The purpose of this study is to show that during and after drinking beer a treatment strategy by insulin bolus and reduction of basal rate reduces the rate of hyperglycaemia without an increase of hypoglycaemic events compared to a treatment strategy according to the standard recommendation without insulin Bolus.

DETAILED DESCRIPTION:
Participants will get two times a height, weight an gender based amount of beer.

One time (Standard) there will be no Insulin given for the beer. Second time (Intervention) half of the carbohydrates containing in the beer will be covered with Insulin, additionally the basal rate will be set to 50% for 12 hours.

All the time, Glucose will be monitored by continuous subcutaneous Glucose Monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participants
* Signed informed consent by parent or legal guardian of adolescent participants <18 years of age
* Age between16-21 years (both including)
* >1 year Type 1 Diabetes
* continuous subcutaneous insulin infusion for at least 3 months
* HbA1c 7-10 % (both including)
* BMI between10-95th percentile for gender and age (both including) for adolescents, <95th percentile for adults
* Ability to wear glucose sensor
* Normal liver enzymes (alanine aminotransferase , aspartate transaminase , Gamma-Glutamyl-Transferase, bilirubin) in age appropriate range by local lab

Exclusion Criteria:

* Severe hypoglycaemia or diabetic ketoacidosis in the past 6 month
* Alcohol or drug abuse
* Psychiatric disorder
* Unstable other metabolic disease as judged by investigator
* Intake of glucocorticoids or growth hormone
* Allergy to adhesive
* Coeliac disease
* Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
• Number of hypoglycaemic events <70 mg/dl per arm from begin of consumption until lunch next day (12:00 am) | 18 hours

SECONDARY OUTCOMES:
• Area under the curve Glucose Sensor >120 mg/dl from begin of drinking to lunch next day | 18 hours
• Total Area under the curve | 18 hours
• average Sensor Glucose from begin of drinking to 12 hours past and to lunch next day | 18 hours
• Time from end of consumption to nadir of serum glucose
• Number of hypoglycaemic events <70 mg/dl per treatment arm until lunch | 18 hours
• Number of hyperglycaemic events > 180 mg/dl per treatment arm until lunch | 18 hours
• Time in Hypoglycaemia <70 mg/dl per treatment arm | 18 hours
• Max. alcohol in expiratory breath | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Torben Biester, MD, Principal Investigator — Study Physician
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krebs HA, Freedland RA, Hems R, Stubbs M. Inhibition of hepatic gluconeogenesis by ethanol. Biochem J. 1969 Mar;112(1):117-24. doi: 10.1042/bj1120117. PMID 5774487
- [Background] Turner BC, Jenkins E, Kerr D, Sherwin RS, Cavan DA. The effect of evening alcohol consumption on next-morning glucose control in type 1 diabetes. Diabetes Care. 2001 Nov;24(11):1888-93. doi: 10.2337/diacare.24.11.1888. PMID 11679452
- [Background] Gin H, Morlat P, Ragnaud JM, Aubertin J. Short-term effect of red wine (consumed during meals) on insulin requirement and glucose tolerance in diabetic patients. Diabetes Care. 1992 Apr;15(4):546-8. doi: 10.2337/diacare.15.4.546. PMID 1499475
- [Background] Jennifer F. Scheel, Karin Schielke, Stefan Lautenbacher, Sabine Aust1, Simone Kremer, Jörg Wolstein; Low-Dose Alcohol Effects on Attention in Adolescents, Zeitschrift für Neuropsychologie, 24 (2), 2013, 103 - 111
- [Background] Koivisto VA, Tulokas S, Toivonen M, Haapa E, Pelkonen R. Alcohol with a meal has no adverse effects on postprandial glucose homeostasis in diabetic patients. Diabetes Care. 1993 Dec;16(12):1612-4. doi: 10.2337/diacare.16.12.1612. PMID 8299457
- [Background] Seidl S, Jensen U, Alt A. The calculation of blood ethanol concentrations in males and females. Int J Legal Med. 2000;114(1-2):71-7. doi: 10.1007/s004140000154. PMID 11197633